CLINICAL TRIAL: NCT05595707
Title: Page 1/27 Effectiveness of an Expert-Guided Early Tracheostomy Pathway for Mechanically Ventilated Critically Ill Adults in Jordan
Brief Title: Expert-Guided Early Tracheostomy Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Denver Health Medical Center (Other)
Responsible Party: Principal Investigator, Ivor Douglas, Professor, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Trachtime22
Record Dates: First submitted 2022-10-09; First posted 2022-10-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Failure; Tracheostomy Complication
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Percutaneous dilatational tracheostomy (Experimental): PDT reccomended for patients with high risk for prolonged mechanical ventilation.
  Interventions: Other: Expert-Guided Early Tracheostomy

INTERVENTIONS:
Other: Expert-Guided Early Tracheostomy — Patients judged to be at moderate to high risk of prolonged ventilation(26, 27) were those who had chronic respiratory failure, advanced Effectiveness of an Expert-Guided Early Tracheostomy Pathway Page 6/27 age, thrombocytopenia or coagulopathy, persistent vasopressor shock, requirement for renal replacement therapy, an admission trauma diagnosis amongst other criteria, were included. In the absence of these criteria, a consensus for low risk of prolonged MV was reached. Early PDT, within the first 7 days from intubation, was recommended for patients with a moderate/high risk of prolonged MV (Early Group). Continued MV by ETT was recommend for low-risk patients with the potential for delayed PDT in the event of delayed weaning and liberation (Late Group).

SUMMARY:
The optimal timing of tracheostomy insertion remains uncertain. We hypothesized that a clinical pathway including expert-informed risk assessment regarding predicted duration of mechanical (MV) would enhance the effectiveness of early percutaneous dilatational tracheostomy (PDT) for patients with anticipated prolonged durations of MV, as reflected by duration of ventilation, complications, and patient-centered outcomes.

DETAILED DESCRIPTION:
three-year prospective observational study (2018-2020) at a tertiary care level 1 trauma center (King Hussein Medical Center) in Amman Jordan and 4 affiliated subspecialty hospitals. The study sequentially enrolled all adult patients (>18yo) with critical illness receiving MV in an intensive care unit for 48 hours or longer. Institutional ethical committee clearance for the study was secured.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing continued MV for 48 or more hours for whom continuation of life-prolonging therapy was indicated

Exclusion Criteria:

Patients at imminent risk of death were included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization from admission to ventilator independent discharge | Hospital stay up to 90 days
  Length of stay in days

SECONDARY OUTCOMES:
Easy or Moderately Easy to Wean | Hospital stay up to 90 days
  Numeric Score
Days of ventilation requiring administration of NMB | Hospital stay up to 90 days
  Fraction of days when patient are mechanically ventilated and received NMB
Difference in average and total morphine equivalent dose | Hospital stay up to 90 days
  Derived dose of morphine equivelants based on potency in mg
90 day survival | 90 days
  Survival recorded through 90 days from admission

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Medical Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No